CLINICAL TRIAL: NCT06656442
Title: "The Effect of Trimetazidine on the Clinical Outcome of Acute Ischemic Stroke Patients"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Tarek Zakaria, Clinical Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMZ and AIS
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stoke; Trimetazidine; metabolic modulator; infarct size; out of window; brain edema; interleukin - 18
MeSH Terms: conditions — Ischemic Stroke; Brain Edema | interventions — Trimetazidine

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, randomized controlled, open-label clinical trial conducted on 60 acute ischemic stroke patients
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trimetazidine and Standard of care (Active Comparator): AIS patients receiving standard of care and Trimetazidine 35mg/12hrs within 12 hours of admission
  Interventions: Drug: Trimetazidine
- Standard of care only (No Intervention): AIS patients receiving standard of care only.

INTERVENTIONS:
Drug: Trimetazidine — an anti-ischemic medication.
  Other Names: Vastarel Mr, Metacardia Mr
  Arms: Trimetazidine and Standard of care

SUMMARY:
The investigators need to test the effect of Trimetazidine on the pro-inflammatory marker Interleukin - 18 , NIHSS score, and mRs score of acute ischemic stroke patients.

DETAILED DESCRIPTION:
Trimetazidine is a well-known anti-anginal drug that exerts its effect by converting the cell's metabolism from fatty acid oxidation to glucose oxidation. This is contrary to what occurs during a stroke event, in which the cell's metabolism is shifted to fatty acid metabolism. It also improves the activity of pyruvate dehydrogenase, the enzyme that allows the entry of pyruvate from the cytosol into the mitochondria for subsequent oxidation in the Krebs cycle. Therefore, attenuating lactic acid production, controlling intracellular acidosis and calcium ion overload, thus conserving valuable ATP stores to meet energy requirements and preventing the occurrence of further ischemia. Clinical reports indicate that trimetazidine restores energy homeostasis and attenuates free radical generation to exhibit benefits in ischemia and angina pectoris.

An increasing number of studies have focused on the effect of Trimetazidine on myocardial I/R injury, and some studies have proposed possible hypotheses. Trimetazidine protects against myocardial I/R injury and is presumed to be related to autophagy, apoptosis, and oxidative stress, which are all pathways in stroke.

An in vitro study proving the role of Trimetazidine in apoptosis found that trimetazidine protected muscle cells against starvation or inflammation-induced atrophy by inhibiting protein degradation and inducing autophagy. It has recently been shown to ameliorate lipopolysaccharide (LPS)-induced cardiomyocyte pyroptosis: which plays an important role in the development of muscle atrophy by promoting neutrophil migration to cardiac tissue. It was shown that Trimetazidine mitigated the mRNA expression of pyroptosis-related molecules, including NLRP3, Caspase-1, and GSDMD.25 In another in vitro study, it was found that TMZ reduced the myocardial infarct size and decreased the expression of TLR4, MyD88, phospho-NF-κB p65, and the NLRP3 inflammasome.

Furthermore, a study assessing the effect of TMZ on cerebral I/R injury proved that it reduced infarct volume compared with the vehicle-treated reperfused animals and significantly decreased the percentage of brain swelling in the TMZ-treated groups.

Trimetazidine in a clinical study added to the standard of care with or without interventional and/or surgical reperfusion reduced oxidative stress, endothelial dysfunction, inflammation, and major acute cardiovascular events, whereas, in patients with chronic coronary syndrome, TMZ decreased oxidative stress and readmission for ACS and heart failure.

Moreover, there is a recent clinical trial that has proven that Trimetazidine significantly reduced the serum levels of interleukin - 18 in patients with acute viral myocarditis compared to the control group.

This makes it possible to detect the severity of the stroke event by measuring the serum levels of interleukin - 18. It is a pro-inflammatory cytokine, that is encoded by the IL-18 gene in humans. It is likely to be the first line of immune defense for the brain, primarily secreted by macrophage cells and mononuclear cells in humans. It is initially expressed as the inactive precursor pro-IL-18. It is then converted into an active form by proteolytic cleavage, mainly by the cysteine protease caspase-1, which is also known as IL-1B converting enzyme (ICE).

Some researchers have proposed the hypothesis that a pro-inflammatory profile induced by increased IL-18 levels creates a prothrombotic and pro-atherosclerotic environment, which may eventually contribute to stroke in older people. These results are consistent with the results of a meta-analysis study which proved that there is a significant association between IL-18 level and NIHSS scores that makes it a strong tool for reflecting the severity of stroke and for predicting the prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) admitted to the stroke unit with a diagnosis of acute ischemic stroke by CT scan after excluding hemorrhagic stroke
* Patients with an NIHSS score between 5 and 25
* Within 6 - 12 hours from the initial symptoms presentation.

Exclusion Criteria:

* Thrombolysis-eligible patients
* Patients already on Trimetazidine for any other indication
* Patients who are NPO
* Patients with impaired liver function are defined as INR of 1.5 or higher, elevated AST and ALT more than 3 times the upper normal limit, thrombocytopenia with platelets, 150, 000 in a patient without cirrhosis or preexisting liver disease.
* Patients with inadequate renal function defined as creatinine clearance of 60 mls/min or less
* Pregnancy and lactation
* Contraindications of trimetazidine such as hypersensitivity to TMZ, Parkinson's disease, tremors, restless leg syndrome, or other movement disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Serum level of interleukin -18 | 7 days
  A decrease in the serum level of the pro-inflammatory marker.
National Institutes of Health Stroke Scale | 7 days
  An improvement in the NIHSS score Minimum: 1 Maximum: 42
The Modified Rankin Score | 90 days
  An improvement in the mRs score Minimum: 0 Maximum: 6
Adverse Effects | Till we reach out sample size: 60 patients (assessed within 1 year)
  Any adverse effect that appeared on the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt